CLINICAL TRIAL: NCT04204785
Title: Noise in the Operating Room at Induction and Patient Satisfaction and Experience (NOISE) Study
Brief Title: Noise in the OR at Induction: Patient and Anesthesiologists Perceptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Trina Montemurro, Clinical Assistant Professor, University of British Columbia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: H19-01798
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Noise Exposure; Surgery; Patient Satisfaction; Anesthesia
Keywords: Operating Room Environment; Noise; General Anesthesia
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Pre-Post Education Survey study
Masking Description: Participants are not randomly assigned to a group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Education (No Intervention): Patient and Anesthesiologist participants completing surveys prior to OR staff education sessions.
- Post-Education (Experimental): Patient and Anesthesiologist participants completing surveys after OR staff education sessions.
  Interventions: Behavioral: Noise Reduction Education

INTERVENTIONS:
Behavioral: Noise Reduction Education — OR staff will be offered education regarding the importance of minimizing noise in the OR. There will also be reminder signs and posters for the duration of the post-education period.
  Arms: Post-Education

SUMMARY:
Noise in the operating room is common and often unavoidable, but there is mixed evidence of its impact. Previous research has suggested that excessive noise at the time when a patient is being 'put to sleep' may lead to care teams missing changes in monitors, having difficulties focusing or increasing stress. However, it is unknown ifs noise at this time affects the patient's satisfaction with the overall surgical experience. The investigators are conducting a survey study to evaluate patients' and anesthesiologists' overall satisfaction at the time of induction, before and after an education program promoting reducing noise in the Operating Room.

Study Purpose: The purpose of this study is to investigate how noise levels that the time of induction in the OR (operating room) effect patient and anesthesiologists' satisfaction with the overall surgical experience.

Hypothesis: The null hypothesis is that there is no improvement in patient satisfaction with the reduction of noise at the time of induction.

Study Population: The Investigators will be including two study populations: patients age 19 or older undergoing elective, non-cardiac surgery with general anesthesia as the primary mode of anesthesia, and; Anesthesiologists working in these rooms.

Research Method: This will be a pre/post survey study of patients and Anesthesiologists perspectives of noise in the OR. The investigators will survey participants before and after an educational intervention for OR staff.

DETAILED DESCRIPTION:
1.0 BACKGROUND: Noise in the operating room (OR) is common whether it be related to surgical equipment, anesthetic monitors, or conversations between health care providers and patients regarding the procedure or patient status. In particular, certain periods can be louder than others, such as during induction and emergence of anesthesia, with preparation and conversations as the major sources of noise during induction. Noise at this time has been shown to lead to deleterious patient outcomes, as staff are unable to hear subtle or even significant changes in monitors, or have difficulty focusing during a critical time of induction. It has also been demonstrated that poor postoperative outcomes in pediatric patients and increase in stress levels in surgeons. While anecdotal, what is not elucidated in the literature is whether or not excess noise during induction affects a patient's perioperative satisfaction. Induction is often a distressing time for patients and extraneous noise may have a significant impact on their overall experience. This study is the first to explore the impact of noise at induction on patient satisfaction investigate whether a reduction in noise on induction can improve patient satisfaction. A secondary outcome is to achieve a decrease in noise level in non-cardiac operating rooms at this facility, promoting the concept of a 'sterile cockpit' (silence during induction) as borrowed from the aviation industry.

2.0 JUSTIFICATION: Studies have demonstrated that excessive noise in the operating room can be associated with critical error. Additionally, it has been shown that for Anesthesiologists' excessive noise can lead to increased. However, the effects of noise in the OR at the time of induction on patient experience remains unclear. While other validated questionnaires regarding patient satisfaction during the perioperative period have been established, these do not include questions regarding noise levels. Thus, this study will be the first to examine how noise during induction will affect patients' perioperative experience.

This tertiary care facility, St. Paul's Hospital, located in Vancouver, British Columbia, does not have a specific protocol or mandate with respect to noise in the operating room at any time. The recommended decibel levels in OR's is <45 decibels.

3.0 STUDY PURPOSE:

The purpose of this study is to:

* Collect data regarding noise levels in the OR at the time of induction
* Collect patient satisfaction survey during phase 1
* Complete noise-reduction strategies (phase 2) to reduce levels of noise in the operating room during the time of induction
* Repeat patient satisfaction survey during phase 3 to determine if patient satisfaction improves with reduction of noise during induction
* Collect data on Anesthesiologist satisfaction survey during phase 1
* Repeat anesthesiologist satisfaction survey during phase 3 to determine if this improves with reduction of noise during induction

4.0 HYPOTHESIS:

The null hypothesis is:

• There is no improvement in patient satisfaction with the reduction of noise at the time of induction.

5.0 OBJECTIVES:

The objectives of this study are to:

* Collect preliminary data regarding noise levels in the OR during induction
* Determine if noise-reduction strategies and education during induction decreases noise levels in the operating room
* Determine if noise-reduction strategies and education improve patient satisfaction in the perioperative period
* Determine if noise-reduction strategies and education improve Anesthesiologist satisfaction during induction

6.0 METHODS & STATISTICS: 6.1 Research Design Overview: Questionnaire Study

This study will take place over three phases.

Phase I:

Measure baseline characteristics of designated non-cardiac, elective operating rooms requiring a general anesthetic as primary mode of anesthesia. This will act as the control group for the study. Data collection will be performed by the attending Anesthesiologist using a portable decibel-meter and a smart phone with a decibel-meter application placed by the patient's head during induction. The Anesthesiologist will use the devices to determine a baseline noise level (maximum and mean decibel levels) in the OR from the time that patient enters the OR to when the patient is successfully intubated. The Anesthesiologist taking the measurement will conceal the devices from the others in the OR (including OR staff and patients). The investigators have received approval from the OR to use this concealed device. The same Anesthesiologist will then fill out a questionnaire regarding patient demographics (e.g. type of procedure, age, anxiety, significant hearing impairment, cognitive impairment) and observed noise in the operating room.

Patient participants will be recruited post-operatively in the postoperative care unit (PACU) and Surgical Day Care (SDC) if they are being discharged home on the same day or on the post-surgical wards if they are being admitted to hospital after surgery. The investigators will recruit patient participants post-operatively so as not to bias their experiences pre-operatively. They will be approached by the perioperative Anesthesiologist when deemed of appropriate mental capacity, to ask if they are willing to hear about the study. If they agree, the perioperative physician will alert a study team member of the eligible patient and they will approach the patient to discuss the study and seek consent. The recruiter will not be involved in the patient's direct care as to ensure patients that their care will not be influenced by whether they decide to participate or not. When recruited, they will complete an anonymous, self-administered questionnaire that will assess their satisfaction or dissatisfaction of care, using a Likert scale questionnaire designed specifically for extraneous noise during the time of induction. A Likert scale questionnaire is used as this has been most validated for perioperative satisfaction in multiple validated questionnaires.

Phase II:

This involves an educational intervention in the form of a didactic teaching session for the surgical teams, Anesthesiologists, Anesthesia Assistants, Perioperative Nurses, and Patient Care Aids The education will be focused on the importance of noise reduction during induction, specifically highlighting its potential positive effects on improving patient outcomes (and potentially patient satisfaction) and impact on surgical teams and Anesthesiologists. This will include formal presentations for each group of OR staff and daily prompts prior to the start of the day slate.

Phase III:

This will be conducted following education of perioperative health care professionals. Exactly the same as phase I, but after education. This involves repeating participant recruitment and data collection, with the Anesthesiologist completing the questionnaire and collecting noise level data, as well as patient participants completing self-administered questionnaires as a repeat of the protocol described above in phase I.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 18 or greater
* Elective, non-cardiac operating room procedure with general anesthesia as the primary mode of anesthesia

Patient Exclusion Criteria:

* Age <19
* Non-elective surgery
* Patients who do not receive General Anesthesia
* Cardiac surgery
* Significant hearing impairment (self-reported)
* Significant cognitive impairment
* Surgeries less than 20 minutes in length
* Medically unstable postoperatively

Anesthesiologist Participants

Anesthesiologist Inclusion Criteria:

* Working in the eligible ORs with eligible patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Change in Maximum Noise Levels Pre-/Post-Education | The time from patient entering the OR to patient being fully intubated ranged from approximately 5 to 20 minutes. The change is measured between the pre- and post-education phases of the study.
  Change in maximum noise levels from pre-education to post-education. Maximum noise levels are measured from the time a patient enters the Operating Room (OR) to the time when the patient is intubated (approximately 5-20 minutes) using an I-phone application (app). The app measures decibel levels and the results were recorded by the anesthesiologist or research assistant.
Change in Average Noise Levels Pre-/Post-Education | The time from patient entering the OR to patient being fully intubated ranged from approximately 5 to 20 minutes. The change is measured between the pre- and post-education phases of the study.
  Change in average/mean noise levels from pre-education to post-education. Mean noise levels are measured from the time a patient enters the Operating Room (OR) to the time when the patient is intubated (approximately 5-20 minutes) using an I-phone application (app). The app measures decibel levels and the results were recorded by the anesthesiologist or research assistant.
Patient Satisfaction Pre-/Post-Education | Patients completed the same surveys in phase 1(pre-education) and phase 3 (post-education). The education was done within a 2 month period after the first phase and before the third phase.
  Patients from the pre-education and post-education groups completed the same satisfaction rating survey. The responses were a combination of yes/no responses and likert scales. The 5-point likert scale response options ranged from: "Strongly disagree, Disagree, Not Sure, Agree, Strongly Agree" and "Not At All, A Little Bit, Moderately, Quite A Bit, Extremely". Responses will be compared between groups by question.

SECONDARY OUTCOMES:
Anesthesiologist Satisfaction Pre-/Post-Education | Anesthesiologists completed the same surveys in phase 1(pre-education) and phase 3 (post-education). The education was done within a 2 month period after the first phase and before the third phase.
  Anesthesiologists completed the same survey in the pre-education and post-education phases. The responses were a combination of yes/no responses, and likert scales. The 5-point likert scale response options ranged from: "Not At All, A Little Bit, Moderately, Quite A Bit, Extremely". Responses will be compared between groups by question.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Katz JD. Noise in the operating room. Anesthesiology. 2014 Oct;121(4):894-8. doi: 10.1097/ALN.0000000000000319. No abstract available. PMID 24878496
- [Background] Ginsberg SH, Pantin E, Kraidin J, Solina A, Panjwani S, Yang G. Noise levels in modern operating rooms during surgery. J Cardiothorac Vasc Anesth. 2013 Jun;27(3):528-30. doi: 10.1053/j.jvca.2012.09.001. Epub 2012 Oct 27. PMID 23107015
- [Background] Hasfeldt D, Laerkner E, Birkelund R. Noise in the operating room--what do we know? A review of the literature. J Perianesth Nurs. 2010 Dec;25(6):380-6. doi: 10.1016/j.jopan.2010.10.001. PMID 21126668
- [Background] Liu EH, Tan S. Patients' perception of sound levels in the surgical suite. J Clin Anesth. 2000 Jun;12(4):298-302. doi: 10.1016/s0952-8180(00)00155-0. PMID 10960202
- [Background] Hogan LJ, Harvey RL. Creating a Culture of Safety by Reducing Noise Levels in the OR. AORN J. 2015 Oct;102(4):410.e1-7. doi: 10.1016/j.aorn.2015.08.005. PMID 26411830
- [Background] Murthy VS, Malhotra SK, Bala I, Raghunathan M. Detrimental effects of noise on anaesthetists. Can J Anaesth. 1995 Jul;42(7):608-11. doi: 10.1007/BF03011878. PMID 7553997
- [Background] Engelmann CR, Neis JP, Kirschbaum C, Grote G, Ure BM. A noise-reduction program in a pediatric operation theatre is associated with surgeon's benefits and a reduced rate of complications: a prospective controlled clinical trial. Ann Surg. 2014 May;259(5):1025-33. doi: 10.1097/SLA.0000000000000253. PMID 24394594
- [Background] Barnett SF, Alagar RK, Grocott MP, Giannaris S, Dick JR, Moonesinghe SR. Patient-satisfaction measures in anesthesia: qualitative systematic review. Anesthesiology. 2013 Aug;119(2):452-78. doi: 10.1097/ALN.0b013e3182976014. PMID 23669268
- [Background] Auquier P, Pernoud N, Bruder N, Simeoni MC, Auffray JP, Colavolpe C, Francois G, Gouin F, Manelli JC, Martin C, Sapin C, Blache JL. Development and validation of a perioperative satisfaction questionnaire. Anesthesiology. 2005 Jun;102(6):1116-23. doi: 10.1097/00000542-200506000-00010. PMID 15915023
- [Background] Caljouw MA, van Beuzekom M, Boer F. Patient's satisfaction with perioperative care: development, validation, and application of a questionnaire. Br J Anaesth. 2008 May;100(5):637-44. doi: 10.1093/bja/aen034. Epub 2008 Mar 12. PMID 18337271
- [Background] Jlala HA, Caljouw MA, Bedforth NM, Hardman JG. Patient satisfaction with perioperative care among patients having orthopedic surgery in a university hospital. Local Reg Anesth. 2010;3:49-55. doi: 10.2147/lra.s11381. Epub 2010 Jul 28. PMID 22915869
- [Background] Mui WC, Chang CM, Cheng KF, Lee TY, Ng KO, Tsao KR, Hwang FM. Development and validation of the questionnaire of satisfaction with perioperative anesthetic care for general and regional anesthesia in Taiwanese patients. Anesthesiology. 2011 May;114(5):1064-75. doi: 10.1097/ALN.0b013e318216e835. PMID 21455058
- [Derived] Yu CV, Foglia J, Yen P, Montemurro T, Schwarz SKW, MacDonell SY. Noise in the operating room during induction of anesthesia: impact of a quality improvement initiative. Can J Anaesth. 2022 Apr;69(4):494-503. doi: 10.1007/s12630-021-02187-9. Epub 2022 Jan 10. PMID 35014000